CLINICAL TRIAL: NCT00837460
Title: Effect of Rehabilitation of Patients With a Central Nervous System Lesion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Fondation Saint Luc (Unknown); Fonds pour la recherche scientifique médicale (FRSM), Belgium (Unknown); Association nationale d'aide aux personnes handicapées (ANAH) (Unknown)
Responsible Party: Cliniques Universitaires Saint-Luc, Université Catholique de Louvain
Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2006/06NOV/207
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Stroke
Keywords: Hand; Rehabilitation
MeSH Terms: conditions — Stroke | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rehabilitation (Experimental): Bilateral and unilateral prehension oriented rehabilitation to enhance prehension.
  Interventions: Other: rehabilitation

INTERVENTIONS:
Other: rehabilitation — 4 weeks of bilateral followed or preceded by 4 weeks of unilateral similar prehension oriented repeated rehabilitation tasks. About 45 minutes 3 times a week, the subject is coached by a physiotherapist to enhance his prehension habilities.

SUMMARY:
The purpose of the study is to analyse the prehensions deficits and the effect of prehension rehabilitation in central nervous system lesioned people

ELIGIBILITY:
Inclusion Criteria:

* Adult minimum 6mounth after first stroke
* Minimal prehension of both hands

Exclusion Criteria:

* Diabetuss
* Other Upper Limb pathologies
* MMSE < 26

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2006-09; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
prehension functionality | 4 weeks before, just before, after first part and after the second part of rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Dispa, PhD student, Principal Investigator — Rehabilitation and physical medecine Unit - UCL; Jean-Louis Thonnard, PhD, Study Director — Rehabilitation and physical medecine Unit-UCL; Yannick Bleyenheuft, PhD student, Principal Investigator — Rehabilitation and physical medecine Unit-UCL; Thierry Lejeune, MD PhD, Study Director — Rehabilitation and physical medecine Unit-UCL
Locations (1):
- READ : Rehabilitation and physical medecine Unit, Brussels, Brussels Capital, Belgium